CLINICAL TRIAL: NCT07352189
Title: Comparison of the Efficacy of Ultrasound-Guided and Laparoscopy-Guided Transversus Abdominis Plane(TAP) Block on Postoperative Analgesia in Patients Undergoing Laparoscopic Upper Abdominal Surgery
Brief Title: Ultrasound-Guided Versus Laparoscopy-Guided Transversus Abdominis Plane Block for Postoperative Analgesia
Acronym: US-LTAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital (Other)
Collaborators: Maltepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MALTEPE-2022-965164
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain Management
Keywords: Transversus Abdominis Plane Block; TAP block; Postoperative Pain; analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided TAP block (Group U) (Experimental): Patients receiving ultrasound-guided subcostal transversus abdominis plane block for postoperative analgesia.
  Interventions: Procedure: Ultrasound-guided Transversus Abdominis Plane (US-TAP) Block
- Laparoscopy-guided TAP block (Group L) (Experimental): Patients receiving laparoscopy-guided transversus abdominis plane block for postoperative analgesia.
  Interventions: Procedure: Laparoscopy-guided Transversus Abdominis Plane (LS-TAP) Block

INTERVENTIONS:
Procedure: Ultrasound-guided Transversus Abdominis Plane (US-TAP) Block — Bilateral ultrasound-guided subcostal transversus abdominis plane block performed prior to extubation using a total of 40 mL local anesthetic solution (30 mL0.25% bupivacaine and 10 ml of 1% lidocaine).
  Arms: Ultrasound-guided TAP block (Group U)
Procedure: Laparoscopy-guided Transversus Abdominis Plane (LS-TAP) Block — Bilateral laparoscopy-guided transversus abdominis plane block performed prior to extubation using a total of 40 mL local anesthetic solution (30 mL 0.25% bupivacaine and 10 ml of 1% lidocaine).
  Arms: Laparoscopy-guided TAP block (Group L)

SUMMARY:
This prospective, randomized, double-blind study aimed to compare the effects of ultrasound-guided versus laparoscopy-guided transversus abdominis plane(TAP) block on postoperative analgesia in patients undergoing laparoscopic upper abdominal surgery under general anesthesia. Postoperative pain scores, analgesic consumption and recovery parameters were evaluated during the first 24 hours after surgery.

DETAILED DESCRIPTION:
Patients aged 18-70 years with ASA physical status I-III who were scheduled for laparoscopic upper abdominal surgery under general anesthesia were included in the study. After induction of anesthesia, patients were randomly assigned to one of two group, bilateral subcostal transversus abdominis plane block was performed under ultrasound-guidance using a local anesthetic mixture before extubation. In the laparoscopy-guided group, bilateral subcostal transversus abdominis plane block was performed under laparoscopic guidance using the same local anesthetic mixture before abdominal closure. Postoperative pain intensity was assessed by using the Numeric Rating Scale (NRS). Total opioid consumption, time to first analgesic requirement, paracetamol consumption, postoperative nausea and vomiting, length of hospital stay, time to ambulation and time to gastrointestinal recovery were recorded during the first 24 hours after surgery. Complications related to the TAP block were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 yeras
* ASA physical status I-III
* Scheduled for laparoscopic upper abdominal surgery
* Provided written informed consent

Exclusion Criteria:

* Patient refusal
* Allergy to local anesthetics
* Coagulopathy
* Infection at the injection site
* Severe systemic disease
* ASA physical status IV-V

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Postoperative pain score (NRS) | First 24 hours postoperatively
  Postoperative pain intensity measured using the Numeric Rating Scale (NRS), a 0-10 scale where 0 indicates no pain and 10 indicates the worst imaginable pain. Higher scores indicates worse pain.

CONTACTS AND LOCATIONS:
Overall Officials: Talat Ercan E Şerifsoy, MD, Principal Investigator — Maltepe University Hospital
Locations (1):
- Maltepe University Faculty of Medicine Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No